CLINICAL TRIAL: NCT00005685
Title: Blood Pressure Control--Racial and Psychosocial Influences
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4131; R01HL031533 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2006-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
To examine racial and psychosocial influences on blood pressure control.

DETAILED DESCRIPTION:
BACKGROUND:

Environmental and psychosocial factors relating to hypertension and cardiovascular disease are incompletely understood, particularly for women and African Americans. Recent research has suggested that job strain is more strongly linked to elevated work blood pressure in men than women. In contrast, the combination of having a high status job plus the trait of high effort coping style (John Henryism) was related to higher work blood pressure in women and African American men, but not Caucasian men.

The grant has been ongoing since September 1983. The original study had as its purpose to ascertain similarities and differences in the etiology of hypertension for Blacks and whites and to identify those biobehavioral factors contributing to the excess risk for hypertension among Blacks. Myocardial, blood pressure, and renal responses (sodium and potassium handling) to laboratory and naturalistic stressors were evaluated in young adult normotensive or marginally hypertensive Black and white men. Behavioral stressors included competitive, reaction time tasks (active coping) as well as more passive coping conditions. Data were collected on family history of hypertension, family social class background, Type A behavior, propensity for anger and hostility, and coping style. The role of the sympathetic nervous system in mediating these effects was assessed by the use of beta-adrenergic antagonists.

When the grant was renewed in 1991, the goal of the research was to evaluate the interactive effects of environmental stressors and sodium chloride (NACl) and potassium (K) intake as they related to hypertension development in a biracial population.

DESIGN NARRATIVE:

There were two studies in the current grant. Study 1 reexamined hypothesized relationships of high effort coping and job strain to elevated ambulatory blood pressure (BP) at work and at home in a sample of 288 Black and white men and women stratified by job status. Also, assessments were made of the relationships of these traits to increased epinephrine and norepinephrine responses, other measures of sympathetic activation, adverse lipid profiles, and cardiac and vascular structural changes. Job strain and high effort coping were also related to hypertension prevalence in 576 black and white men and women stratified by job status. The influence of additional psychosocial variables (social support, hostility, anger-in, depressed mood, anxiety) was also examined.

Study 2 built on prior research on gender differences in total peripheral resistance during stressors which enhance alpha-adrenergic activity, and on a recent observation that among young adults, slow sodium excretion during stress is seen in five times as many men as women. It also built on recent work suggesting that estrogen may attenuate total peripheral resistance responses to stress by reducing vasoconstrictive effects of alpha-adrenergic activity. The study was designed to examine cardiovascular, lipid, epinephrine, norepinephrine, and sodium excretion responses to stressors in 120 subjects maintained for a week on a controlled high salt diet. Thirty subjects were tested in each of these groups: 1) premenopausal women, 2) postmenopausal women not using hormone replacement therapy, 3) postmenopausal women using hormone replacement, 4) men. Each group included 15 Black and 15 white subjects, and each subject was tested twice, once after receiving placebo and once after receiving either an alpha- or a beta-receptor antagonist.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1983-09; Study Completion 2002-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Light — University of North Carolina

REFERENCES:
- [Background] Girdler SS, Turner JR, Sherwood A, Light KC. Gender differences in blood pressure control during a variety of behavioral stressors. Psychosom Med. 1990 Sep-Oct;52(5):571-91. doi: 10.1097/00006842-199009000-00009. PMID 2247562
- [Background] Turner JR, Sherwood A. Postural effects on blood pressure reactivity: implications for studies of laboratory-field generalization. J Psychosom Res. 1991;35(2-3):289-95. doi: 10.1016/0022-3999(91)90083-z. PMID 2046061
- [Background] Hinderliter AL, Light KC, Willis PW 4th. Left ventricular mass index and diastolic filling. Relation to blood pressure and demographic variables in a healthy biracial sample. Am J Hypertens. 1991 Jul;4(7 Pt 1):579-85. doi: 10.1093/ajh/4.7.579. PMID 1873012
- [Background] Turner JR, Sherwood A, Light KC. Generalization of cardiovascular response: supportive evidence for the reactivity hypothesis. Int J Psychophysiol. 1991 Aug;11(2):207-12. doi: 10.1016/0167-8760(91)90013-n. PMID 1748596
- [Background] Hinderliter AL, Light KC, Willis PW 4th. Gender differences in left ventricular structure and function in young adults with normal or marginally elevated blood pressure. Am J Hypertens. 1992 Jan;5(1):32-6. doi: 10.1093/ajh/5.1.32. PMID 1736932
- [Background] Light KC, Turner JR. Stress-induced changes in the rate of sodium excretion in healthy black and white men. J Psychosom Res. 1992 Jul;36(5):497-508. doi: 10.1016/0022-3999(92)90011-p. PMID 1619590
- [Background] Light KC, Turner JR, Hinderliter AL. Job strain and ambulatory work blood pressure in healthy young men and women. Hypertension. 1992 Aug;20(2):214-8. doi: 10.1161/01.hyp.20.2.214. PMID 1639463
- [Background] Sherwood A, Royal SA, Hutcheson JS, Turner JR. Comparison of impedance cardiographic measurements using band and spot electrodes. Psychophysiology. 1992 Nov;29(6):734-41. doi: 10.1111/j.1469-8986.1992.tb02051.x. PMID 1461960
- [Background] Light KC, Dolan CA, Davis MR, Sherwood A. Cardiovascular responses to an active coping challenge as predictors of blood pressure patterns 10 to 15 years later. Psychosom Med. 1992 Mar-Apr;54(2):217-30. doi: 10.1097/00006842-199203000-00007. PMID 1565757
- [Background] Girdler SS, Hinderliter AL, Light KC. Peripheral adrenergic receptor contributions to cardiovascular reactivity: influence of race and gender. J Psychosom Res. 1993;37(2):177-93. doi: 10.1016/0022-3999(93)90085-t. PMID 8385216
- [Background] Sherwood A, Hinderliter AL. Responsiveness to alpha- and beta-adrenergic receptor agonists. Effects of race in borderline hypertensive compared to normotensive men. Am J Hypertens. 1993 Jul;6(7 Pt 1):630-5. doi: 10.1093/ajh/6.7.630. PMID 8398005
- [Background] Light KC, Turner JR, Hinderliter AL, Sherwood A. Race and gender comparisons: I. Hemodynamic responses to a series of stressors. Health Psychol. 1993 Sep;12(5):354-65. doi: 10.1037//0278-6133.12.5.354. PMID 8223359
- [Background] Light KC, Turner JR, Hinderliter AL, Sherwood A. Race and gender comparisons: II. Predictions of work blood pressure from laboratory baseline and cardiovascular reactivity measures. Health Psychol. 1993 Sep;12(5):366-75. doi: 10.1037//0278-6133.12.5.366. PMID 8223360
- [Background] Turner JR, Sherwood A, Light KC. Intertask consistency of hemodynamic responses to laboratory stressors in a biracial sample of men and women. Int J Psychophysiol. 1994 Jul;17(2):159-64. doi: 10.1016/0167-8760(94)90031-0. PMID 7995778
- [Background] Hinderliter AL, Light KC, Willis PW 4th. Patients with borderline elevated blood pressure have enhanced left ventricular contractility. Am J Hypertens. 1995 Oct;8(10 Pt 1):1040-5. doi: 10.1016/0895-7061(95)00256-1. PMID 8845073
- [Background] Hinderliter AL, Sager AR, Sherwood A, Light KC, Girdler SS, Willis PW 4th. Ethnic differences in forearm vasodilator capacity. Am J Cardiol. 1996 Jul 15;78(2):208-11. doi: 10.1016/s0002-9149(96)90397-5. PMID 8712144
- [Background] Light KC, Brownley KA, Turner JR, Hinderliter AL, Girdler SS, Sherwood A, Anderson NB. Job status and high-effort coping influence work blood pressure in women and blacks. Hypertension. 1995 Apr;25(4 Pt 1):554-9. doi: 10.1161/01.hyp.25.4.554. PMID 7721397
- [Background] Sherwood A, Hinderliter AL, Light KC. Physiological determinants of hyperreactivity to stress in borderline hypertension. Hypertension. 1995 Mar;25(3):384-90. doi: 10.1161/01.hyp.25.3.384. PMID 7875764
- [Background] Brownley KA, Light KC, Anderson NB. Social support and hostility interact to influence clinic, work, and home blood pressure in black and white men and women. Psychophysiology. 1996 Jul;33(4):434-45. doi: 10.1111/j.1469-8986.1996.tb01069.x. PMID 8753944
- [Background] Brownley KA, West SG, Hinderliter AL, Light KC. Acute aerobic exercise reduces ambulatory blood pressure in borderline hypertensive men and women. Am J Hypertens. 1996 Mar;9(3):200-6. doi: 10.1016/0895-7061(95)00335-5. PMID 8695017
- [Background] Girdler SS, Pedersen CA, Light KC. Thyroid axis function during the menstrual cycle in women with premenstrual syndrome. Psychoneuroendocrinology. 1995;20(4):395-403. doi: 10.1016/0306-4530(94)00068-9. PMID 8532823
- [Background] Light KC, Girdler SS, Sherwood A, Bragdon EE, Brownley KA, West SG, Hinderliter AL. High stress responsivity predicts later blood pressure only in combination with positive family history and high life stress. Hypertension. 1999 Jun;33(6):1458-64. doi: 10.1161/01.hyp.33.6.1458. PMID 10373233
- [Background] West SG, Light KC, Hinderliter AL, Stanwyck CL, Bragdon EE, Brownley KA. Potassium supplementation induces beneficial cardiovascular changes during rest and stress in salt sensitive individuals. Health Psychol. 1999 May;18(3):229-40. doi: 10.1037//0278-6133.18.3.229. PMID 10357504
- [Background] West SG, Brownley KA, Light KC. Postexercise vasodilatation reduces diastolic blood pressure responses to stress. Ann Behav Med. 1998 Spring;20(2):77-83. doi: 10.1007/BF02884452. PMID 9989312
- [Background] Brownley KA, Hinderliter AL, West SG, Girdler SS, Sherwood A, Light KC. Sympathoadrenergic mechanisms in reduced hemodynamic stress responses after exercise. Med Sci Sports Exerc. 2003 Jun;35(6):978-86. doi: 10.1249/01.MSS.0000069335.12756.1B. PMID 12783046
- [Background] Grewen KM, Girdler SS, Hinderliter A, Light KC. Depressive symptoms are related to higher ambulatory blood pressure in people with a family history of hypertension. Psychosom Med. 2004 Jan-Feb;66(1):9-16. doi: 10.1097/01.psy.0000106881.60228.16. PMID 14747632